CLINICAL TRIAL: NCT02214953
Title: An Open, Randomised, Single-dose, Four-way Cross-over Formulation Finding Study of the Oral Bioavailability of Four Prototype Extended Release Formulations With 25 mg BI 11634, and Intra-individual Comparison to Immediate-release Tablets (25 mg) in Healthy Male Volunteers
Brief Title: Bioavailability of Four Oral Prototype Extended Release Formulations With BI 11634 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1234.7
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (5):
- BI 11634 ER formulation A (Experimental)
  Interventions: Drug: BI 11634 ER formulation A
- BI 11634 ER formulation B (Experimental)
  Interventions: Drug: BI 11634 ER formulation B
- BI 11634 ER formulation M (Experimental)
  Interventions: Drug: BI 11634 ER formulation M
- BI 11634 ER formulation C (Experimental)
  Interventions: Drug: BI 11634 ER formulation C
- BI 11634 IR tablet (Active Comparator)
  Interventions: Drug: BI 11634 IR tablet

INTERVENTIONS:
Drug: BI 11634 ER formulation A
  Arms: BI 11634 ER formulation A
Drug: BI 11634 ER formulation B
  Arms: BI 11634 ER formulation B
Drug: BI 11634 ER formulation M
  Arms: BI 11634 ER formulation M
Drug: BI 11634 ER formulation C
  Arms: BI 11634 ER formulation C
Drug: BI 11634 IR tablet
  Arms: BI 11634 IR tablet

SUMMARY:
To compare the oral bioavailability and rate of absorption of four prototype extended-release (ER) formulations with BI 11634 (single doses) to immediate-release (IR) tablets in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian males according to the following criteria, based upon a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate), 12-lead ECG, clinical laboratory tests
* Age ≥21 and ≤45 years
* Haemoglobin within the normal ranges.
* Body Mass Index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and the local legislation

Exclusion Criteria:

* Relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Relevant surgery of gastrointestinal tract
* History of any bleeding disorder or acute blood coagulation defect, for the subject itself or any person of his family as far as known
* History of gastric ulcera and cholecystectomy
* Occult blood in faeces
* Relevant diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Relevant chronic or acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Use of acetylsalicylic acid or any other non-steroidal anti-inflammatory drugs (NSAID) within 2 weeks of study start until the end of study
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Alcohol abuse (more than 40 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to understand and comply with protocol requirements, instructions and protocol stated restrictions, the nature, scope and possible consequences of the study
* Subjects with a history within the past six weeks of closed-head or torso trauma or deceleration injury such as an automobile accident or fall from a significant height

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 48 hours after drug administraton
Cmax (maximum measured concentration of analyte in plasma) | up to 48 hours after drug administraton

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 48 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 48 hours after drug administration
λz (terminal rate constant in plasma) | up to 48 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 48 hours after drug administration
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 48 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 48 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 48 hours after drug administration
Fluctuation parameter Cmax/C24 ratio | up to 48 hours after drug administration
Maximum prolongation of blood coagulation time | up to 48 hours after drug administration
  by HepTest® (Haemachem Inc.)
Number of subjects with adverse events | up to 8 days after last drug administration
Number of subjects with clinically significant findings in vital signs (blood pressure, pulse rate) | up to 8 days after last drug administration
Number of subjects with clinically significant findings in ECG | up to 8 days after last drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 8 days after last drug administration
Assessment of tolerability by investigator on a 4-point scale | up to 8 days after last drug administration
% Inhibition of Factor Xa | up to 48 hours after drug administration
  by Russel's Viper Venom test (RVV)